CLINICAL TRIAL: NCT03350633
Title: Safety and Efficacy of Tocilizumab Versus Azathioprine in Neuromyelitis Optica Spectrum Disorders: a Randomized, Controlled, Open-label, Phase 2 Trial
Brief Title: Tocilizumab vs Azathioprine in Neuromyelitis Optica Spectrum Disorders
Acronym: TANGO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Director of Neurology Department, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-YX-009
Record Dates: First submitted 2017-11-10; First posted 2017-11-22 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica | interventions — tocilizumab; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab Injection (ACTEMRA®) , a IL-6 receptor blockade
  Interventions: Drug: Tocilizumab Injection
- Azathioprine (Active Comparator): Imuran
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Tocilizumab Injection — Tocilizumab Injection will be intravenously administered with a dose of 8 mg/kg every 4 weeks.
  Other Names: ACTEMRA®
  Arms: Tocilizumab
Drug: Azathioprine — Azathioprine will be orally given at a dose of 2-3 mg/kg/d
  Other Names: Imuran
  Arms: Azathioprine

SUMMARY:
In neuromyelitis optica spectrum disorder (NMOSD),interleukin-6 (IL-6) may play an important role in facilitating plasma cells to produce pathological aquaporin 4 (AQP4) autoantibody. Inhibition of IL-6 signaling pathway by Tocilizumab (ACTEMRA®), a humanized monoclonal antibody may have shown beneficial clinical effects in a few patients with NMOSD.

Larger scale clincial trials may be needed to observe its efficacy and safety. Here, by choosing azathioprine, one of the most frequently used medication in case of relapses, the investigators compare the safety and efficacy of tocilizumab in preventing NMOSD attacks.

DETAILED DESCRIPTION:
The investigators primarily aim to observe the time to first relapse from initiation of tocilizumab or azathioprine treatment. The proportion of participants who experience relapse-free in one year follow-up will be compared.

The secondary outcomes are to determine: The safety profile of tocilizumab and azathioprine in participants with NMO and whether tocilizumab improves visual function, Expanded Disability Status Scale (EDSS), et al.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old
2. Diagnosis of NMO or NMO spectrum disorder
3. Clinical evidence of at least 2 relapses in last 12 months or 3 relapses in the last 24 months
4. Able and willing to give written informed consent and comply with the requirements of the study protocol.
5. EDSS <= 7.5 (8 in special circumstances)
6. Men and women of reproductive potential must agree to use a highly effective method of birth control from screening to 6 months after final dose of the investigational product.

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection (Herpes simplex virus, varicella-zoster virus, cytomegalovirus, Epstein-Barr virus,human immunodeficiency virus, Hepatitis viruses, Syphilis, etc)
2. Pregnant, breastfeeding, or child-bearing potential during the course of the study
3. Patients will not participate in any other clinical therapeutic study or will not have participated in any other experimental treatment study within 30 days of screening
4. Participation in another interventional trial within the last 3 months
5. Heart or kidney insufficiency
6. Tumor disease currently or within last 5 years
7. Clinically relevant liver, kidney or bone marrow function disorder
8. Intolerance of azathioprine or previous relapses on azathioprine treatment
9. Receipt of rituximab or any experimental B-cell depleting agent within 6 months prior screening and B-cells below the lower limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Time to first relapse | From baseline to one year after
  An acute attack was defined as a new neurological worsening lasting for at least 24 hours and occurring more than 30 days after the previous attack.

SECONDARY OUTCOMES:
Proportion of patients who experience relapse-free | From baseline to 60 weeks
  To record whether the patients had no relapses in the follow-ups
Worsening in EDSS | Worsening from baseline in EDSS to 60 weeks
  The Expanded Disability Status Scale (EDSS) is a rating system that is frequently used for classifying and standardizing the severity and progression. EDSS ranges from 0 to 10.
Time to Onset of Confirmed Disability Progression (CDP) for at Least 12 Weeks | From baseline to 60 weeks
  Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening. Participants who had initial disability progression with no confirmatory EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Percentage of Participants With Confirmed Disability Improvement (CDI) for at Least 12 Weeks | From baseline to 60 weeks
  Disability improvement was assessed only for the subgroup of participants with a baseline EDSS score of >= 2.0. It was defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was >=2 and <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death).
Time to Onset of Confirmed Disability Progression (CDP) for at Least 24 Weeks | From baseline to 60 weeks
  Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death). Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. Participants who had initial disability progression with no confirmatory EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Percentage of Participants With Confirmed Disability Improvement (CDI) for at Least 24 Weeks | From baseline to 60 weeks
  Disability improvement was assessed only for the subgroup of participants with a baseline EDSS score of >= 2.0. It was defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was >=2 and <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death).
Percentage Change in Spectral-domain Optical Coherence Tomography (SD-OCT) Average Retinal Nerve Fiber Layer (RNFL) Thickness at Week 60 | From baseline to 60 weeks
  Adjusted mean percentage change in thickness of the RNFL at Week 60 for the affected eye from the baseline as determined by SD-OCT.
Percentage change in SD-OCT Average Retinal Ganglion Cell Layer/Inner Plexiform Retinal Layer (RGCL/IPL) at Week 60 | From baseline to 60 weeks
  Adjusted mean change in thicknesses of the RGCL/IPL at Week 60 for the affected eye from the baseline as determined by segmentation of SD-OCT.
Change in Low-contrast Letter Acuity (LCLA) at Week 60 | From baseline to 60 weeks
  Adjusted mean change in LCLA at Week 60 from baseline as determined by 2.5% low contrast Sloan letter charts, adjusted for the baseline LCLA value.
Change in High-contrast Letter Acuity (HCLA) at Week 60 | From baseline to 60 weeks
  Adjusted mean change in HCLA at Week 60 from baseline as determined by 100% high contrast Sloan letter charts, adjusted for the baseline HCLA value.
Number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Brain Magnetic Resonance Imaging (MRI) | From baseline to 60 weeks
  The total number of new and/or enlarging T2 lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 12, 36, and 60
Overall safety and tolerability of tocilizumab or azathioprine | From baseline to 60 weeks
  Adverse events related to tocilizumab or azathioprine are recorded.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From baseline to 60 weeks
  Treatment-emergent adverse events, treatment-emergent serious adverse events (TESAEs), including laboratory measurements as well as their changes or shift from baseline over time
Counts of peripheral blood B cell subsets | From baseline to 60 weeks
  Compare peripheral blood plasma cells before and one year after initial intervention
Determination of serum immunoglobulins | From baseline to 60 weeks
  Compare immunoglobulins before and one year after initial intervention
Determination of serum AQP4 antibodies | From baseline to 60 weeks
  Compare serum AQP4-ab titers before and one year after initial intervention
Determination of serum cytokines | From baseline to 60 weeks
  Compare serum cytokines before and one year after initial intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang C, Zhang M, Qiu W, Ma H, Zhang X, Zhu Z, Yang CS, Jia D, Zhang TX, Yuan M, Feng Y, Yang L, Lu W, Yu C, Bennett JL, Shi FD; TANGO Study Investigators. Safety and efficacy of tocilizumab versus azathioprine in highly relapsing neuromyelitis optica spectrum disorder (TANGO): an open-label, multicentre, randomised, phase 2 trial. Lancet Neurol. 2020 May;19(5):391-401. doi: 10.1016/S1474-4422(20)30070-3. PMID 32333897